CLINICAL TRIAL: NCT02846805
Title: A Clinical Trial on Conventional Dentures and Implant-retained Mandibular Overdentures With Respect to Oral Functionality and Quality of Life in Edentulous Patients
Brief Title: The Treatment of Implant-retained Mandibular Overdentures for Edentulous Patients
Acronym: TIMOEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chufan Ma (Other)
Responsible Party: Sponsor-Investigator, Chufan Ma, Associate professor, Air Force Military Medical University, China
Organization: Air Force Military Medical University, China (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-REV-2016035
Record Dates: First submitted 2016-07-03; First posted 2016-07-27 (Estimated); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Edentulous
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- complete dentures (No Intervention): complete dentures will be provided for all subjects according to the standardized treatment protocol
- implant-retained overdentures (Experimental): subjects will receive two-implant-retained overdentures in the mandible ,and continue wearing their complete denture in the maxilla
  Interventions: Procedure: implant-retained overdentures

INTERVENTIONS:
Procedure: implant-retained overdentures — subjects will receive two-implant-retained overdentures in the mandible,and they continue wearing their complete denture in the maxilla.
  Arms: implant-retained overdentures

SUMMARY:
The purpose of this study is to investigate to what extent IOs improve the functionality of edentulous patients and changes in quality of life and overall patient satisfaction following treatment with IOs.

DETAILED DESCRIPTION:
Edentulous individuals will be selected from patients attending the prosthodontic clinic. Then, new complete dentures will be provided; in a second stage half of these subjects (randomly selected) will receive IOs. The effect of different treatment protocols on chewing ability, patient satisfaction and OHRQoL will be investigated and assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Being edentulous in the upper and lower jaw for at least 1 year
2. Dissatisfied or cannot function with their complete lower denture
3. Age between 40 and 75
4. Suitable bone quality as assessed radiographically (CBCT) according to Zarb's classification。

Exclusion Criteria:

1. Physical and mental disabilities which interfere with the maintenance of implants;
2. Severe skeletal jaw discrepancies (class III)
3. Those who have already received or lost dental implants
4. Those who abuse drugs or alcohol
5. Smoking more than 10 cigarettes a day
6. Having received radiotherapy to the head and neck region for malignancies
7. Undergoing chemotherapy
8. On long-term therapy with steroids
9. immunosuppressants or biphosphonates
10. Insulin-dependent diabetic patients and uncontrolled onset diabetic patients
11. Those affected by chronic renal or liver disease
12. Systemic and local bone disorders and pathology
13. Serious cardiac and pulmonary disorders
14. Haemophilic disorders who are susceptible for increased bleeding and tendency for post-operative infections
15. Those who are at risk of developing bacterial endocarditis
16. Immune system compromised patients, including those with HIV

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
masticatory efficiency | three months after restoration of the implant-retained overdenture
  masticatory efficiency will be measured with chwing-gum ,and the outcome will be analysed with the viewgum software

SECONDARY OUTCOMES:
Oral health related quality of life | three months after restoration of the implant-retained overdenture
  Oral health related quality of life will be measured with the Oral Health Impact Profile 14(OHIP-14).
patients' satisfaction | three months after restoration of the implant-retained overdenture
  patients' satisfaction will be assessed on visual analog scales (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Chufan Ma, Study Chair — Air Force Military Medical University, China
Locations (1):
- Department of Prosthodontics,School of Stomatology,The Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No
secret